CLINICAL TRIAL: NCT02425995
Title: Prevalence and Diagnosis of Hidden Lesions of the Posterior Horn of the Medial Meniscus in Pediatric Anterior Cruciate Ligament (ACL) Lesions : Interest of Arthroscopic Intercondylar and Posteromedial Portals
Brief Title: Interest of Additional Arthroscopic Portals in Diagnosis of Hidden Lesions of the Medial Meniscus in Pediatrics Knees With ACL Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL14_0358
Record Dates: First submitted 2015-04-15; First posted 2015-04-24 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Knee Instability
Keywords: ACL; Hidden lesions of the medial meniscus; Chronic knee instability; Intercondylar and posteromedial arthroscopy; Arthroscopic Posteromedial and Intercondylar portal; Diagnosis capacity of hidden lesions of the medial meniscus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arthroscopic intercondylar and posteromedial portal (Experimental)
  Interventions: Procedure: Arthroscopic intercondylar and posteromedial portal

INTERVENTIONS:
Procedure: Arthroscopic intercondylar and posteromedial portal — Diagnosis of lesions of the Posterior Horn of the Medial Meniscus in Arthroscopic intercondylar and posteromedial portal in addition with standard ACL reconstruction, during the same surgery.

SUMMARY:
Peroperatively observative study in pediatric orthopedic center in Lyon, France.

50 pediatric patients included in this study, to improve the diagnosis of hidden lesions of the medial meniscus associated with lesions of the anterior cruciate ligament.

All the patients need a reconstruction of the ACL because of chronic knee instability.

All the patients underwent a multi portal arthroscopy during the ACL reconstruction : anteromedial and anterolateral and after intercondylar and posteromedial.

The study consists in a peroperatively arthroscopic look, in order to diagnose lesions of the posterior horn of the medial meniscus which could be missed in MRI and anteromedial and anterolateral arthroscopy.

Statistics of this lesions are used to study prevalence and diagnosis capacity of this procedures.

First, the surgeon did a classic knee arthroscopy. Secondarily, he did an intercondylar portal and after a posteromedial portal.

ELIGIBILITY:
Inclusion Criteria:

- Chronic knee instability with indicated surgery reconstruction

Exclusion Criteria:

* Pregnancy
* No preoperatively knee MRI
* Posteromedial or Intercondylar Portal Failure
* Social security system membership failure
* Refusal of consent of child or parents

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of hidden lesions diagnosed in Arthroscopic Posteromedial Portal and not seen in classic arthroscopic portals and Intercondylar Portal. | Day 1 (during surgery)
  Diagnosis of a hidden lesion of the Posterior Horn of the Medial Meniscus in Arthroscopic Posteromedial Portal, which has not be seen in classic arthroscopic portals and Intercondylar Portal.

SECONDARY OUTCOMES:
Number of hidden lesions diagnosed during the arthroscopic procedure and not seen in preoperatively MRI. | Day 1 (during surgery)
  Diagnosis of a hidden lesion of the posterior horn of the medial meniscus during the arthroscopic procedure, lesion not seen in preoperatively MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Franck CHOTEL, Pr, Principal Investigator — Service de Chirurgie Orthopédique Pédiatrique - Hôpital Femme Mère Enfant - 59, Bd Pinel 69677 BRON CEDEX
Locations (1):
- Hospices Civils de Lyon, Lyon, France